CLINICAL TRIAL: NCT01792934
Title: A Randomized Multicenter Clinical Trial for Patient With Multi-organ, Colorectal Cancer Metastases Comparing the Combination of Chemotherapy and Maximal Tumor Debulking Versus Chemotherapy Alone.
Brief Title: Chemotherapy and Maximal Tumor Debulking of Multi-organ Colorectal Cancer Metastases
Acronym: ORCHESTRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-073
Record Dates: First submitted 2012-12-20; First posted 2013-02-15 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Multi-organ Metastatic Colorectal Cancer
Keywords: Debulking, cytoreduction, RFA, SABR, palliative chemotherapy
MeSH Terms: interventions — Surgical Procedures, Operative; Radiofrequency Ablation; Radiosurgery; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX or FOLFOX regimen (Active Comparator): XELOX or FOLFOX regimen
  Interventions: Drug: XELOX regimen according to standard procedures; Drug: FOLFOX regimen according to standard procedures; Drug: Bevacizumab; Procedure: tumor biopsy
- XELOX or FOLFOX regimen and maximal tumor debulking (Experimental): XELOX or FOLFOX regimen and maximal tumor debulking including Surgery, radiofrequency ablation (RFA), transarterial chemo-embolization using irinotecan drug-eluted beads ((DEBIRI)-TACE) or stereotactic body radiation therapy (SBRT).
  Interventions: Drug: XELOX regimen according to standard procedures; Drug: FOLFOX regimen according to standard procedures; Procedure: Surgery; Other: radiofrequency ablation (RFA); Other: transarterial chemo-embolization using irinotecan drug-eluted beads ((DEBIRI-)TACE); Radiation: stereotactic body radiation therapy (SBRT); Drug: Bevacizumab; Procedure: tumor biopsy

INTERVENTIONS:
Drug: XELOX regimen according to standard procedures
Drug: FOLFOX regimen according to standard procedures
Procedure: Surgery
  Arms: XELOX or FOLFOX regimen and maximal tumor debulking
Other: radiofrequency ablation (RFA)
  Arms: XELOX or FOLFOX regimen and maximal tumor debulking
Other: transarterial chemo-embolization using irinotecan drug-eluted beads ((DEBIRI-)TACE)
  Arms: XELOX or FOLFOX regimen and maximal tumor debulking
Radiation: stereotactic body radiation therapy (SBRT)
  Arms: XELOX or FOLFOX regimen and maximal tumor debulking
Drug: Bevacizumab — may be added to both regimens according to standard procedures
Procedure: tumor biopsy — at baseline (diagnostic or study) biopsy and after 3 or 4 cycles an optional tumor biopsy

SUMMARY:
The purpose of this study is to compare overall survival rates of colorectal cancer patients with multi-organ metastases with an indication for first line systemic treatment randomized for treatment with combination chemotherapy or treatment with combination chemotherapy and additional maximal tumor debulking including surgical tumor resection, RFA, (DEBIRI-)TACE and SBRT, depending on best clinical judgement according to a standardized treatment algorithm. Our hypothesis is that maximal tumor debulking in addition to systemic treatment with chemotherapy and biologicals will provide an improvement in progression free and overall survival in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of cancer is required.
* Indication for first line palliative systemic treatment for metastatic colorectal cancer (mCRC).
* Patients with CRC metastases in (the primary tumor is excluded as metastatic site)

  * ≥ 2 different organs if at least >1 extra-hepatic metastases or
  * ≥ 2 different organs including >5 hepatic metastases not located to one lobe or
  * ≥ 2 different organs including either a positive para-aortal lymph nodes or celiac lymph nodes or adrenal metastases or pleural carcinomatosis or peritoneal carcinomatosis
* Feasible radical tumor debulking. Incomplete tumor debulking is allowed only if at least 80% of metastases can be treated.
* To meet the inclusion criteria a cytological analysis should be performed in case of any uncertainty about the presence of a lesion e.g. a false positive or false negative result on imaging.
* Age ≥ 18 years.
* WHO performance status 0 - 1.
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin ≥ 5.6 mmol/L;
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3;
  * Platelet count ≥ 100*109/l;
  * Total bilirubin ≤ 1.5 times the upper limit of normal;
  * ALT and AST ≤ 2.5 x upper limit of normal (≤ 5 x upper limit of normal for subjects with liver involvement of their cancer);
  * Albumin > 30 g/l;
  * Serum creatinine ≤ 1.5 x upper limit of normal or a MDRD ≥ 50 ml/min;
  * Prothrombin time or INR < 1.5 x ULN, unless coumarin derivates are used. Due to interactions with capecitabine, all patients using coumarin derivates will be treated with LMWH instead.
  * Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed if this treatment can be interrupted as judged by the treating physician).
* Written informed consent.

Exclusion Criteria:

* Prior (neo-)adjuvant chemotherapy for < 6 months after last treatment and first detection of extra-hepatic metastases, except for neoadjuvant capecitabine in the context of chemoradiation for rectal carcinoma.
* Candidates for HIPEC.
* Patients with liver metastases only
* Evidence of brain metastases.
* History of other prior malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Patients with other malignancies are eligible if they have remained disease free for at least 5 years.- History of cardiac disease:

  * Congestive heart failure >NYHA class 2;
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening);
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mm Hg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 3 separate measurements on at least 2 separate days.
* Uncontrolled infections (> grade 2 NCI-CTC version 4.0).
* Pregnant or breast-feeding women. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g., cervical cap, condom, and diaphragm) or intrauterine device during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised.
* Concurrent anticancer chemotherapy, immunotherapy or investigational drug therapy during the study or within 4 weeks of the start of study drug.
* Concomitant use of dexamethasone, anticonvulsants and anti-arrhythmic drugs other than digoxin or beta blockers.
* Severe allergy for contrast media not controlled with premedication.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from date of study inclusion until the date of death or until the end of follow up, assessed up to 10 years

SECONDARY OUTCOMES:
Progression free survival rates | date of study inclusion to the first event defined as local recurrence or progression, distant recurrence or death from any cause assessed up to 10 years
Response rates | assessed every 3 months, after a follow up of 3 years assessed every 6 months
Safety and efficacy of the additional local treatment measured by number of serious adverse events. | assessed after inclusion of 25, 50 and 100 patients, after 30% of the patients are included in the study for 12 months and after the end of follow up, assessed up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: H.M.W. Verheul, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (29):
- Netherlands (27):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuis Groep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Amstelveen Ziekenhuis, Amstelveen
  - VU Medical Center, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Gelre, Apeldoorn
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Albert Schweizer ziekenhuis, Dordrecht
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Hospital, Flushing
  - Dijklander, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Radboud University Medical Center, Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Erasmus University Medical Center, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - IJsselland ziekenhuis, Rotterdam
  - Maasstadziekenhuis, Rotterdam
  - Medisch Centrum Haaglanden, The Hague
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - Zaans Medisch Centrum, Zaandam
  - Isala Klinieken, Zwolle
- United Kingdom (2):
  - University College London Hospital, London
  - University Hospital Southampton, Southampton

REFERENCES:
- [Derived] Bakkerus L, Buffart LM, Buffart TE, Meyer YM, Zonderhuis BM, Haasbeek CJA, Versteeg KS, Loosveld OJL, de Groot JWB, Hendriks MP, Verhoef C, Verheul HMW, Gootjes EC. Health-Related Quality of Life in Patients With Metastatic Colorectal Cancer Undergoing Systemic Therapy With or Without Maximal Tumor Debulking. J Natl Compr Canc Netw. 2023 Oct;21(10):1059-1066.e5. doi: 10.6004/jnccn.2023.7050. PMID 37856212